CLINICAL TRIAL: NCT04372108
Title: An Observational Study to Assess the Long-term Safety of Ustekinumab Versus Other Biologic Therapies Among Patients With Crohn's Disease and Ulcerative Colitis: A New-User Cohort Study Using the Department of Defense Electronic Health Records Database
Brief Title: A Study to Assess the Long-Term Safety of Ustekinumab Versus Other Biologics in Patients With Crohn's Disease and Ulcerative Colitis
Status: Recruiting | Type: Observational
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108561; RRA-18896 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-04-30; First posted 2020-05-01 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Crohn Disease; Colitis, Ulcerative
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative | interventions — Ustekinumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ustekinumab New User Cohort: Participants with crohn's disease (CD) or ulcerative colitis (UC) with no prior exposure to ustekinumab, at least 1 year of enrollment records immediately prior to the new use will be required. The information will be sourced from the Department of Defense (DoD) Electronic Health Records (EHR) database in the United States (US).
  Interventions: Drug: Ustekinumab
- Other Biologics Comparator Cohort: Participants with CD or UC with no prior exposure to the individual drugs (for example, infliximab, adalimumab, or vedolizumab) in question, at least 1 year of enrollment records immediately prior to the new use of the comparator biologic will be required. The information will be sourced from the Department of Defense (DoD) Electronic Health Records (EHR) database in the United States (US).
  Interventions: Drug: Other Biologic Therapies

INTERVENTIONS:
Drug: Ustekinumab — Participants who are new users of ustekunumab will be included in the cohort. No study treatment will be administered as a part of this study.
  Groups: Ustekinumab New User Cohort
Drug: Other Biologic Therapies — Participants who are new users of other biologic therapies (for examples for example, infliximab, adalimumab, or vedolizumab administered as per the prescription record) will be included in this cohort. No study treatment will be administered as a part of this study.
  Groups: Other Biologics Comparator Cohort

SUMMARY:
The purpose of this study is to estimate and compare the incidence of overall malignancy, serious infection, and opportunistic infections between new users of ustekinumab and new users of other biologic therapies among adult participants with Crohn's disease (CD) or ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women with CD or UC who are new users of ustekinumab or the comparator drugs during the study period
* Participants must have at least 1 year of enrollment history with the DoD EHR database immediately prior to new use (that is, exposure index date) of ustekinumab or the comparator drugs

Exclusion Criteria:

* Participants below 18 years of age on the exposure index date
* Participants who do not meet the definition for CD or UC prior to or on the exposure index date
* Participants with any records of human immunodeficiency virus (HIV) diagnosis, organ or tissue transplant, or malignancy (excluding non-melanoma skin cancer [NMSC]) at any time prior to or on the exposure index date
* Participants with a physician diagnosis of rheumatoid arthritis, ankylosing spondylitis, or psoriatic arthritis within 12 months prior to or on the exposure index date
* In the analysis of infection outcomes, participants diagnosed with the same infection of interest both within 60 days prior to or on the exposure index date and within 60 days after the exposure index date will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include participants with Crohn's Disease (CD) or Ulcerative Colitis (UC) who are new users of ustekinumab and new users of the comparator drugs which will be identified from the Department of Defense (DoD) Electronic Health Records (EHR) database.
Sampling Method: Probability Sample
Enrollment: 1056 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2030-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence Rate for Malignancy | Up to 10 years and 3 months
  The incidence rates for malignancy (including Non-melanoma skin cancer [NMSC]) will be estimated as the number of incident cases (that is, counts of unique participants) divided by the total at-risk time.

SECONDARY OUTCOMES:
Opportunistic Infection (OI) | Up to 10 years and 3 months
  The OI will be estimated as the number of incident cases (that is counts of unique participants) divided by the total at-risk time.
Serious Infection | Up to 10 years and 3 months
  The serious infections will be estimated as the number of incident cases (that is counts of unique participants) divided by the total at-risk time.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (1):
- NMCP, Portsmouth, Virginia, United States